CLINICAL TRIAL: NCT02206022
Title: REMIFENTANIL AND LOCAL ANESTHESIA COMPARED WITH LOCAL ANESTHESIA FOR THE INSERTION OF CENTRAL VENOUS CATHETERS IN AWAKE PATIENTS
Brief Title: Remifentanil And Local Anesthesia Compared With Local Anesthesia For The Insertion Of Central Venous Catheters
Acronym: REMIDOLCATH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13 6932 03
Record Dates: First submitted 2014-03-10; First posted 2014-08-01 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Local Anesthesia
Keywords: Central Venous Catheter; Remifentanil; local anesthesia; pain
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Experimental): Patients who undergone a Central Venous Catheter (CVC) insertion under remifentanil infusion
  Interventions: Drug: Remifentanil
- Placebo (Placebo Comparator): Patients who undergone a Central Venous Catheter (CVC) insertion under placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remifentanil — Pain's evaluation for Remifentanil Group
  Arms: Remifentanil
Drug: Placebo — CVC pain's evaluation after local anesthesia + placebo infusion
  Arms: Placebo

SUMMARY:
At present, there is no reference protocol for Central Venous Catheter (CVC) insertion assuring analgesia, anxiolysis and safety. Medical teams use various levels of analgesia and anesthesia to realize this gesture, from single local anesthesia to general anesthesia. Remifentanil has been shown to decrease pain scores for insertion and removal of long-term central venous access. Remifentanil is also often employed for pediatric or labor analgesia for short acts as procedural sedation.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* eligible for CVC insertion

Exclusion Criteria:

* pregnancy
* patients who can't give their consent
* contra-indications to remifentanil infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Maximal pain score on numeric rating scale (NRS) will be assessed after the insertion | up to 60 minutes

SECONDARY OUTCOMES:
Evaluation of patient's anxiety by the Face Anxiety Scale | up to 60 minutes
Patient and physician's satisfaction by a 10-points numeric rating scale | up to 60 minutes
Number of adverse events | up to 60 minutes
Number of realized punctions | up to 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean RUIZ, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vardon Bounes F, Pichon X, Ducos G, Ruiz J, Samier C, Silva S, Sommet A, Fourcade O, Conil JM, Minville V. Remifentanil for Procedural Sedation and Analgesia in Central Venous Catheter Insertion: A Randomized, Controlled Trial. Clin J Pain. 2019 Aug;35(8):691-695. doi: 10.1097/AJP.0000000000000725. PMID 31094935